CLINICAL TRIAL: NCT04417816
Title: Ultrasound-induced Adipose Tissue Cavitation: Effects on Cardiometabolic Risk and Body Composition in Persons With Obesity
Brief Title: Ultrasound-induced Adipose Tissue Cavitation and Training in Obesity
Acronym: UATC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the request of the Ethical Committee
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UATC-001
Record Dates: First submitted 2020-05-15; First posted 2020-06-05 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training + adipose tissue cavitation (Experimental)
  Interventions: Other: Exercise training intervention with ultrasound induced adipose tissue cavitation
- Exercise training + sham procedure (Sham Comparator)
  Interventions: Other: Exercise training intervention without ultrasound induced adipose tissue cavitation

INTERVENTIONS:
Other: Exercise training intervention with ultrasound induced adipose tissue cavitation — Exercise training intervention with ultrasound induced adipose tissue cavitation
  Arms: Exercise training + adipose tissue cavitation
Other: Exercise training intervention without ultrasound induced adipose tissue cavitation — Exercise training intervention with ultrasound induced adipose tissue cavitation
  Arms: Exercise training + sham procedure

SUMMARY:
The addition of ultrasound-induced adipose tissue cavitation (UATC) at the level of the abdominal subcutaneous adipose tissue may seem relevant as an additive treatment option to exercise intervention in individuals with obesity. However, whether individuals with obesity who participate in an exercise intervention and additionally undergo UATC, are more likely to develop a metabolically healthy phenotype, as opposed to subjects with obesity undergoing exercise training or UATC only, remains to be studied. Therefore, the first aim of this study is to examine the impact of combined UATC during exercise intervention on abdominal subcutaneous and whole-body adipose tissue mass, quality of life and cardiometabolic risk in individuals with abdominal obesity.

ELIGIBILITY:
Inclusion Criteria:

* male/female (1:1),
* age 18-65 y,
* abdominal obesity (waist circumference >102cm or >88cm) -

Exclusion Criteria:

* involvement in dietary or exercise intervention in the last year,
* intake of any medication,
* clinically diagnosed diseases (cardiovascular disease, hypertension, venous thromboses blood diseases, presence of a pacemaker/defibrillator, brain or nervous system diseases, kidney, thyroid or liver disease, chronic inflammatory diseases, cancer, osteoporosis and epilepsy).
* Persons with a pregnancy,
* a recent bone injury or the presence of a metal prothese

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
DEXA scan | baseline
  Body composition (fat mass, fat free mass, android and gynoid fat mass), clinical measures (waist circumference, hip circumference, weight, height)
DEXA scan | week 12
  Body composition (fat mass, fat free mass, android and gynoid fat mass), clinical measures (waist circumference, hip circumference, weight, height)
Fasting blood sample | Baseline
  (glycated haemoglobin)
Fasting blood sample | week 12
  (glycated haemoglobin)
lipid profile | Baseline
  total LDL, HDL, triglycerides
lipid profile | week 12
  total LDL, HDL, triglycerides
kidney function | Baseline
  urea, creatinine
kidney function | week 12
  urea, creatinine
inflammation | Baseline
  CRP
inflammation | week 12
  CRP
Bloodpressure | Baseline
  systolic and diastolic blood pressure
Bloodpressure | Week 12
  systolic and diastolic blood pressure
oral glucose tolerance test | Baseline
  glucose and insulin levels at 0, 15, 30, 45, 60, 90 and 120 min post glucose load
oral glucose tolerance test | week 12
  glucose and insulin levels at 0, 15, 30, 45, 60, 90 and 120 min post glucose load

SECONDARY OUTCOMES:
Overall physical fitness | Baseline
  Maximal oxygen uptake (during cardiopulmonary exercise testing)
Overall physical fitness | week 12
  Maximal oxygen uptake (during cardiopulmonary exercise testing)
Overall physical fitness | Baseline
  Maximal resistance (during cardiopulmonary exercise testing)
Overall physical fitness | week 12
  Maximal resistance (during cardiopulmonary exercise testing)
Overall physical fitness | Baseline
  Maximal heart rate (measured by electrocardiogram)
Overall physical fitness | week 12
  Maximal heart rate (measured by electrocardiogram)
SF-36 questionaire | Baseline
  Quality of Life questionaire, a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status
SF-36 questionaire | week 12
  Quality of Life questionaire, a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status
Food intake | Baseline
  3-day food diary
Food intake | week 12
  3-day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University; Kenneth Verboven, dr., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Belgium